CLINICAL TRIAL: NCT01304823
Title: The Role of Sweet Taste Receptor Blockade on Intraduodenal Glucose- and Liquid Meal-stimulated Secretion of Satiation Peptides in Healthy Humans
Brief Title: Role of the Gut Sweet Taste Receptor in the Secretion of Glucagon-like Peptide-1 and Peptide YY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EKBB 69/04.03
Record Dates: First submitted 2011-02-22; First posted 2011-02-25 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Taste Disorder, Primary, Sweet
Keywords: T1R2/T1R3; gastric emptying; gut; lactisole; nutrient sensing
MeSH Terms: conditions — Taste Disorders | interventions — lactisole; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- glucose (Active Comparator): intraduodenal perfusion of glucose (29.3 g glucose per 100 mL; rate: 2.5 mL/min for 180 min; caloric load: 3.0 kcal/min)
  Interventions: Dietary Supplement: lactisole
- glucose + lactisole (Active Comparator): intraduodenal perfusion of glucose (29.3 g glucose per 100 mL; rate: 2.5 mL/min for 180 min; caloric load: 3.0 kcal/min) + 450 ppm lactisole
  Interventions: Dietary Supplement: lactisole
- mixed liquid meal (Active Comparator): intraduodenal perfusion of a mixed liquid meal (20.20 g carbohydrate, 4.92 g fat and 6.25 g protein per 100 mL; rate: 2.5 mL/min for 180 min; caloric load: 3.0 kcal/min)
  Interventions: Other: mixed liquid meal
- mixed liquid meal + lactisole (Active Comparator): intraduodenal perfusion of a mixed liquid meal (20.20 g carbohydrate, 4.92 g fat and 6.25 g protein per 100 mL; rate: 2.5 mL/min for 180 min; caloric load: 3.0 kcal/min) + 450 ppm lactisole
  Interventions: Other: mixed liquid meal
- saline + lactisole (Placebo Comparator): saline (0.9 %; rate: 2.5 mL/min for 180 min) + 450 ppm lactisole
  Interventions: Dietary Supplement: lactisole

INTERVENTIONS:
Dietary Supplement: lactisole — flavoring agent/sweet taste antagonist
  Other Names: Dietary supplement
  Arms: glucose; glucose + lactisole; saline + lactisole
Other: mixed liquid meal — Ensure Plus
  Other Names: Dietary supplement
  Arms: mixed liquid meal; mixed liquid meal + lactisole

SUMMARY:
The purpose of this study is to determine the functional significance of sweet taste receptors in the secretion of GI satiation peptides by using a specific sweet taste receptor antagonist to block sweet taste perception in the gastrointestinal tract.

DETAILED DESCRIPTION:
There is strong evidence that taste signaling mechanisms identified in the oral epithelium also operate in the gut. It is suggested that open-type enteroendocrine cells directly sense nutrient via alpha-gustducin coupled taste receptors to modulate the secretion of glucagon like peptide-1 (GLP-1) and peptide YY (PYY). Several nutrient responsive G-protein coupled receptors have been identified in the human gut, including the sweet taste responsive T1R2/T1R3 heterodimer, the amino acid/umami responsive T1R1/T1R3 as well as GPR120 for unsaturated long-chain free fatty acids.The functional significance of sweet taste receptors in the secretion of GLP-1 and PYY will be determined by intraduodenal perfusion of glucose (I) or a mixed liquid meal (II) with or without lactisole (450 ppm) in a double blind, 5-way crossover trial including 10 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* BMI of 19.0-24.5
* Age 18-40
* stable body weight for at least 3 month

Exclusion Criteria:

* smoking
* substance abuse
* regular intake of medication
* medical or psychiatric illness
* gastrointestinal disorders or food allergies

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal peptide secretion | 4 hours blood sampling
  Assessment of venous GLP-1 and PYY release to meal stimulation with and without sweet receptor blockade

SECONDARY OUTCOMES:
Appetite perceptions during 4 hours using VAS | 4 hours
  Assessment of the following appetite perception markers: feelings of hunger, feelings of fullness, feelings of satiety using validated visual analogue scales

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — Phase 1 Research Unit, University Hospital Basel
Locations (1):
- University Hospital Basel, Phase 1 Research Unit, Basel, Switzerland

REFERENCES:
- [Result] Steinert RE, Meyer-Gerspach AC, Beglinger C. The role of the stomach in the control of appetite and the secretion of satiation peptides. Am J Physiol Endocrinol Metab. 2012 Mar 15;302(6):E666-73. doi: 10.1152/ajpendo.00457.2011. Epub 2012 Jan 3. PMID 22215654
- [Result] Steinert RE, Gerspach AC, Gutmann H, Asarian L, Drewe J, Beglinger C. The functional involvement of gut-expressed sweet taste receptors in glucose-stimulated secretion of glucagon-like peptide-1 (GLP-1) and peptide YY (PYY). Clin Nutr. 2011 Aug;30(4):524-32. doi: 10.1016/j.clnu.2011.01.007. Epub 2011 Feb 15. PMID 21324568